CLINICAL TRIAL: NCT04680234
Title: Comparative Study Between the Effect of Superficial Cryotherapy Using Dimethyl Ether and Propane Mixture and Microneedling in Treatment of Alopecia Areata
Brief Title: Superficial Cryotherapy Versus Microneedling in Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zeinab Abu elbaha Gouda, Assistant lecturer of Dermatology, Venereology and Andrology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alopecia2020
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Alopecia Areata
Keywords: alopecia areata; Microneedling; Cryotherapy
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups (randomly assigned and comparably cross matched for age and sex) Cryotherapy group (No.= 50): Superficial cryotherapy using dimethyl ether and propane (DMEP) at -57C Microneedling group (No. = 50): Microneedling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryotherapy group (Active Comparator): Patients underwent superficial cryotherapy using dimethyl ether and propane (DMEP) at -57C very 2 weeks for maximum six sessions
  Interventions: Procedure: DMEP kit
- Microneedling group (Active Comparator): Patients underwent microneedling 2 weeks for maximum six sessions
  Interventions: Device: Dermapen

INTERVENTIONS:
Procedure: DMEP kit — Superficial Cryotherapy using dimethyl ether and propane (DMEP) at -57C
  Arms: Cryotherapy group
Device: Dermapen — Under aseptic precautions, the dermapen was moved on the alopecic patches diagonally, vertically and horizontally 4 to 5 times in each direction Pin point bleeding was taken as an end point
  Arms: Microneedling group

SUMMARY:
This study is randomized comparative analytical prospective study that included patients with mild and moderate alopecia areata. Patients was divided into two groups Patients in the first group underwent Superficial cryotherapy using dimethyl ether and propane (DMEP) at -57C (Cryotherapy group). Patients in the second group underwent Microneedling (Microneedling group). A total of six sessions were done at 2 weeks interval. Patients were followed-up for next 3 months to evaluate the persistence of hair regrowth after therapy. Patients were assessed at baseline and during follow up using photography, Dermoscopy, SALT score and regrowth scale.

ELIGIBILITY:
Inclusion Criteria:

* ِAlopecia areata patients

Exclusion Criteria:

* Alopecia totalis and universalis
* ِAge less than four years.
* ِPregnancy or breast-feeding.
* ِActive infection at the site alopecia patch(s).
* ِInflammation ate site of the alopecia patches
* ِIntolerance to cold.
* ِAssociated systemic illness such as thyroid, pernicious anaemia, diabetes mellitus, autoimmune connective tissue diseases.
* ِPrevious treatment for alopecia areata over the last three months.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Regrowth Scale | Change in regrowth scale from baseline to 3 months follow after end of sessions
  0 score (regrowth < 10%) no response
  1. score (regrowth 11-25%) poor response
  2. score (regrowth 26-50%) fair response
  3. score (regrowth 51-75%) satisfactory response
  4. score (regrowth ≥ 75%) excellent response.

SECONDARY OUTCOMES:
SALT score | Change in salt score from baseline to 3 months follow after end of sessions
  SALT score is the sum of the percentage of hair loss in all the abovementioned areas. For example, if the percentage hair loss in vertex, right profile, left profile, and posterior aspect is 20, 30, 40, and 50% respectively; then, SALT score = (20 × 0.4) = (30 × 0.18) + (40 × 0.18) + (50 × 0.24) = 8 + 5.4 + 7.2 + 12 = 32.6.

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab A Gouda, MSc, Study Director — Sohag Faculty of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data will be provided upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Always
Access Criteria: Request to prinicipal investigator